CLINICAL TRIAL: NCT03728348
Title: An Evaluation of a Multi-target Stool DNA (Mt-sDNA) Test, Cologuard, for CRC Screening in Individuals Aged 45-49 and at Average Risk for Development of Colorectal Cancer: Act Now
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-10
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Cancer
Keywords: Sample Collection; Stool DNA; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual stool samples may be used to develop and evaluate the performance of biomarker assays to detect cancers. Sample may be stored for up to 20 years. These stool samples will be de-identified.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subject aged 45-49 with Average CRC Risk: Subject aged 45-49 with average risk for development of CRC.
  Interventions: Diagnostic Test: mt-sDNA screening test; Procedure: Colonoscopy

INTERVENTIONS:
Diagnostic Test: mt-sDNA screening test — Stool samples will be collected by the subject for the mt-sDNA screening test.
  Other Names: Cologuard
Procedure: Colonoscopy — Subjects will undergo a screening colonoscopy.

SUMMARY:
The primary objective is to confirm the specificity of a multi-target stool DNA test (mt-sDNA), Cologuard, in an average risk population, ages 45-49.

DETAILED DESCRIPTION:
Subjects aged 45-49 at average risk for development of CRC will be enrolled. Subjects will complete the mt-sDNA screening test (Cologuard) followed by completion of a screening colonoscopy. The results of the mt-sDNA screening test (Cologuard) will not be provided to investigators for clinical management of study subjects. Personnel performing the colonoscopy and producing the resulting report and personnel performing histopathological review of tissue (if applicable) will remain blinded to the results of the mt-sDNA screening test (Cologuard) result.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria to be eligible for the study:

1. Subject is at average risk for development of CRC.
2. Subject is able and willing to undergo a screening colonoscopy.
3. Subject is ≥ 45 and ≤ 49 years of age at the time of enrollment.
4. Subject is willing and able to sign informed consent.
5. Subject is able and willing to provide stool sample(s) according to written instructions provided.

Exclusion Criteria:

1. Subject has a history of CRC or adenoma.
2. Subject has ≥2 first-degree relatives who have been diagnosed with CRC
3. Subject has one first-degree relative with CRC diagnosed before the age of 60.
4. Subject has any of the following: Overt rectal bleeding, e.g., hematochezia or melena within the previous 30 days (blood on toilet paper, after wiping, does not constitute rectal bleeding). Positive fecal occult blood test or FIT within the previous six (6) months. Subject has had a previous colonoscopy. Subject has undergone any double-contrast barium enema, virtual (CT-based) colonoscopy, or flexible sigmoidoscopy within the previous five (5) years.
5. Subject has a diagnosis or personal history of any of the following conditions, including: Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP and Gardner's syndrome). Hereditary non-polyposis CRC syndrome (also referred to as "HNPCC" or "Lynch Syndrome").Other hereditary cancer syndromes including but are not limited to Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Neurofibromatosis and Familial Hyperplastic Polyposis.
6. Subject has a family history of: Familial adenomatous polyposis (also referred to as "FAP"), Hereditary non-polyposis CRC syndrome (also referred to as "HNPCC" or "Lynch Syndrome").
7. Subjects with Cronkhite-Canada Syndrome.
8. Subject has a diagnosis of inflammatory bowel disease (IBD) including chronic ulcerative colitis (CUC) and Crohn's disease.
9. Subject has a history of aerodigestive tract cancer.
10. Subject has had a prior colorectal resection for any reason other than sigmoid diverticular disease.
11. Subject has any condition that in the opinion of the investigator should preclude participation in the study.

Ages: 45 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects 45-49 years of age who are at average risk for development of CRC. 942 subjects are targeted to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 983 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Imperiale, MD, Principal Investigator — Indiana University
Locations (39):
- United States (39):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Ventura County Gastroenterology, Camarillo, California
  - Alliance Research Centers, Laguna Hills, California
  - Focilmed, Oxnard, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Yale University Section of Digestive Diseases and Liver Diseases, New Haven, Connecticut
  - Precision Clinical Research, LLC, Lauderdale Lakes, Florida
  - Northshore University Health System Evanston Hospital, Evanston, Illinois
  - DM Clinical Research- Southwest Gastroenterology, Oak Lawn, Illinois
  - Deaconess Clinic- Mt. Pleasant, Evansville, Indiana
  - Indiana University, Eskanazi Hospital, Indianapolis, Indiana
  - Deaconess Clinic- Gateway, Newburgh, Indiana
  - Johnson County ClinTrials, LLC, Lenexa, Kansas
  - New Orleans Research Institute, Metairie, Louisiana
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - Investigative Clinical Research, Annapolis, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - Capitol Research, Rockville, Maryland
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - United Medical Associates, Binghamton, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - Charlotte Gastroenterology & Hepatology, PLLC, Charlotte, North Carolina
  - Wilmington Gastroenterology Associates, Wilmington, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Family Practice Center of Wooster, Inc./Clinical Trial Developers, Massillon, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Comprehensive Internal Medicine, Inc., Wooster, Ohio
  - Gastroenterology Associates, PA, Greenville, South Carolina
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - University of Texas Health Science Center- McGovern Medical School, Houston, Texas
  - DM Clinical Research- PCP for Life, Houston, Texas
  - Virginia Gastroenterology Institute, Suffolk, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after de-identification. This may include text, tables, figures, and appendices. The study protocol, statistical analysis plan, informed consent form, and clinical study report will also be shared. Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available from 2 years and ending 4 years after publication.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research.

REFERENCES:
- [Derived] Imperiale TF, Kisiel JB, Itzkowitz SH, Scheu B, Duimstra EK, Statz S, Berger BM, Limburg PJ. Specificity of the Multi-Target Stool DNA Test for Colorectal Cancer Screening in Average-Risk 45-49 Year-Olds: A Cross-Sectional Study. Cancer Prev Res (Phila). 2021 Apr;14(4):489-496. doi: 10.1158/1940-6207.CAPR-20-0294. Epub 2021 Jan 12. PMID 33436397

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 983 participants provided written informed consent.
Groups:
- Average Risk Patients: Subjects were men and women 45-49 years of age, inclusive, who were at average risk of developing colorectal cancer. We compared results of a noninvasive, multitarget stool DNA test to colonoscopy. Histopathology was performed on any biopsy or excised lesions.
Period: Overall Study
Arm/Group | Average Risk Patients
Started | 983
Did Not Complete Study Procedures | 107
Multi-target DNA Test Excluded | 15
Colonoscopy Excluded | 19
Completed | 842
Not Completed | 141

BASELINE CHARACTERISTICS:
Population: All evaluable participants except for participants who had mt-sDNA or colonoscopy excluded.
Groups:
- Average Risk Patients: Subjects were men and women 45-49 years of age, inclusive, who were at average risk of developing colorectal cancer. We compared results of a noninvasive, multi-target stool DNA test to colonoscopy. Histopathology was performed on any biopsy or excised lesions.
Arm/Group | Average Risk Patients
Number analyzed (Participants) | 842
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 402
  Male | 440
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 48
  Ethnicity: Not Hispanic or Latino | 794
  Race: White | 706
  Race: Black or African American | 95
  Race: Asian | 31
  Race: American Indian or Alaska Native | 1
  Race: Native Hawaiian or Other Pacific Islander | 1
  Race: Other | 8
Region of Enrollment [Number; unit: participants]
  United States | 842
BMI: mean (SD) [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (5.9)
Cigarette Smoking History n(%) [Count of Participants; unit: Participants]
  Never Smoked | 582
  Former Smoker | 174
  Current Smoker | 86

OUTCOME MEASURES:

1. Primary Outcome: Specificity of the Multi-target Stool DNA Test in Average Risk Population, Ages 45-49
Description: An optical colonoscopic procedure is the reference method. Lesions will be confirmed as malignant by histopathologic examination. Results were generated with the use of a logistic-regression algorithm, with values of 183 or more considered to be positive. Tests were processed independently of colonoscopic findings. The test functions as a screening tool by generating a score, based on the detection of hemoglobin and multiple DNA methylation and mutational markers, together with an assessment of the total amount of human DNA in each sample. Specificity =100*(multi-target stool DNA test negative/negative colonoscopy)
Time Frame: Through study completion, an average of 60 days
Population: All completed participants that had a negative colonoscopy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Multi-target DNA Test Results: Subjects were men and women 45-49 years of age, inclusive, who were at average risk of developing colorectal cancer. We compared results of a noninvasive, multitarget stool DNA test to colonoscopy. Histopathology was performed on any biopsy or excised lesions.
Arm/Group | Multi-target DNA Test Results
Number analyzed (Participants) | 792
percentage of participants | 95.3 [93.6 to 96.7]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 60 days
Description: Only device related adverse events were collected.
Arm/Group | Average Risk Patients
All-Cause Mortality (participants affected / at risk) | 0/983
Serious Adverse Events (participants affected / at risk) | 0/983
Other Adverse Events (participants affected / at risk) | 0/983

LIMITATIONS AND CAVEATS:
Subjects with colonoscopic non-advanced adenoma findings were included in the specificity analysis as disease status negative. The colonoscopically 'negative' population included subjects with no findings on colonoscopy and have a higher specificity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator agreed that they shall not, without the Sponsor's prior written consent, independently publish, publicly disclose, present or discuss any results of or information pertaining to the activities conducted under their agreement for a period of one (1) year following completion of the Study.

DOCUMENTS (3):
  • Study Protocol: Version 2 (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT03728348/Prot_000.pdf
  • Study Protocol: Version 1 (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT03728348/Prot_001.pdf
  • Statistical Analysis Plan (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT03728348/SAP_002.pdf